CLINICAL TRIAL: NCT00079612
Title: Randomized Discontinuation Study of BAY 43-9006 in Patients With Advanced Refractory Cancer.
Brief Title: Study of Nexavar (Sorafenib, BAY 43-9006) in Patients With Advanced Refractory Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100391; NCT00044499 (obsolete NCT alias)
Record Dates: First submitted 2004-03-09; First posted 2004-03-11 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Cancer; RCC; Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — 800mg daily (2x 400mg tabs)
  Arms: Arm 1
Drug: Placebo — 2x 400mg tabs daily
  Arms: Arm 2

SUMMARY:
The purpose of the study is to:

* Find out if BAY 43-9006 prevents the growth of tumors
* For patients who have stable cancer status after 3 months of treatment if it is safer and/or more effective to continue to give BAY 43-9006 or to stop giving BAY 43-9006 at that time.
* Find out how long the effect of BAY 43-9006 is on tumors. To assess the safety of BAY 43-9006 (sorafenib) in the treatment of advanced refractory cancers.
* Measure the amount of BAY 43-9006 and some of its targets in the blood stream in some patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years- Patients with refractory solid cancer for which curative or palliative measures have failed or patients whose treatments are considered ineffective or intolerable
* Patients with non-colorectal cancers are eligible and must be progressing at the time of the screening assessment and for whom no other treatment exists
* Patients with at least one (1) measurable tumor, per the WHO Tumor Response Criteria - Histological or cytological documentation of cancer- ECOG Performance status 0 or 1
* Life expectancy of at least 12 weeks- Adequate bone marrow, liver and renal function (assessed by the following laboratory requirements):
* Hemoglobin >/= 9.0 g/dl - Absolute neutrophil count (ANC) >/=1,500/mm3
* Platelet count = 100,000/µl3
* Total bilirubin </=1.0 times the upper limit of normal unless due to Gilbert's
* ALT and AST </= 2.5 x upper limit of normal. (For patients with hepatic involvement of their cancer, ALT and AST < 5.0 x upper limit of normal)
* PT-INR/PTT < 1.5 x upper limit of normal. (Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.

In addition, these patients must be monitored with weekly coagulation assessments throughout the Run-in Period)- Serum creatinine < 1.5 x upper limit of normal

Exclusion Criteria:

* Patients who meet the following criteria at the time of screening will be excluded:
* Non small cell lung cancer, hepatocellular cancer, CML and AML
* Serious cardiac arrhythmia
* Congestive Heart Failure (NYHA Class 3 or 4)
* Active of coronary artery disease or ischemia
* Active acute infections that could be worsened by anticancer therapy or interfere with this study
* Known HIV infection
* Metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry
* Patients currently receiving medication (steroid or anticonvulsant therapy) for seizure disorder
* History of organ allograft- Previous or concurrent cancer that is distinct from the cancer being evaluated in this study. Several situations are excluded, including cervical carcinoma in situ, adequately treated basal cell carcinoma, superficial bladder tumors or any cancer definitively treated greater than 3 years
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to the first dose of study drug
* Radiotherapy during the study or within 3 weeks prior to the first dose of study drug
* Bone marrow transplant or stem cell rescue within 4 months prior to the first dose of study drug
* Biological response modifiers, such as G-CSF within 3 weeks prior to study entry
* Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study
* Investigational drug therapy outside of this trial during or within 4 weeks prior to the screening assessment
* Any previous exposure to a Ras pathway inhibitor
* Pregnant or breast feeding patients. Women of child bearing potential must have a negative pregnancy test. Adequate barrier contraception will be required for both male and female patients during the entire course of the trial
* Substance abuse, medical or psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with the trial
* Any condition that is unstable or could jeopardize the safety of the patient and/or their compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2002-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Number of progressions post randomization to placebo or sorafenib | 12 weeks post randomization

SECONDARY OUTCOMES:
Time to progression | Until Progression occurs
Duration of objective tumor response | Time from initial Response to documented Tumor Progression
Overall survival time | At the End-of-Study visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (4):
  - Chicago, Illinois
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
- United Kingdom (3):
  - London, Greater London
  - Glasgow, Strathclyde
  - Sutton, Surrey

REFERENCES:
- See also: #PL#PubMed. — http://www.ncbi.nlm.nih.gov/pubmed/16636341?dopt=AbstractPlus